CLINICAL TRIAL: NCT01214629
Title: A Phase I Study of LY2523355 in Patients With Advanced Cancer
Brief Title: A Study for Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11618; I1Y-MC-JFBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Advanced Cancer; Metastatic Cancer; Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — litronesib; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2523355 (Experimental)
  Interventions: Drug: LY2523355
- LY2523355 + pegfilgrastim (Experimental)
  Interventions: Drug: LY2523355; Drug: pegfilgrastim

INTERVENTIONS:
Drug: LY2523355 — Administered intravenously as a 1-hour infusion on Days 1, 2, 3 of each 21-day cycle for at least 2 cycles. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion is met. Starting dose for LY2523355 alone arm is 0.125 milligrams per meter square per day (mg/m²/day).
  Arms: LY2523355
Drug: LY2523355 — Administered intravenously as a 1-hour infusion on Days 1, 2, 3 of each 21-day cycle for at least 2 cycles. Participants may continue on study drug until disease progression, unacceptable toxicity or other withdrawal criterion is met. Starting dose for LY2523355 + pegfilgrastim is 4 mg/m²/day.
  Arms: LY2523355 + pegfilgrastim
Drug: pegfilgrastim — 6 milligrams (mg) administered subcutaneously on Day 4 of each 21-day cycle for the 2 planned cycles and for any subsequent cycles of LY2523355 received.
  Arms: LY2523355 + pegfilgrastim

SUMMARY:
This study is being conducted to determine the safety of LY2523355 for the treatment of advanced and/or metastatic cancer (including Non-Hodgkin's lymphoma).

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized, open label, dose-escalation, Phase 1 study of intravenous LY2523355 in participants with advanced and/or metastatic cancer (including Non-Hodgkin's Lymphoma) for whom no treatment of higher priority exists.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of advanced and/or metastatic cancer (solid tumors or Non-Hodgkin's lymphoma) that is refractory to standard therapy or for which no proven effective therapy exists. Participants entering Part B of the study must also have a tumor that is safely amenable to serial biopsies
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST, Therasse et al. 2000) or Revised International Working Group Lymphoma Response Criteria (Cheson et al. 2007)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 28 days (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with child bearing potential must have had a negative urine or serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Have an estimated life expectancy of greater than or equal to 12 weeks

Exclusion Criteria:

* Have symptomatic, untreated or uncontrolled central nervous system (CNS) metastases. Participants with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic participants without history of CNS metastases is not required
* Have current acute or chronic leukemia
* Have had an autologous or allogenic bone marrow transplant
* Have the following conduction abnormalities: PR >250 milliseconds (msec), second degree or complete atrioventricular (AV) block, intraventricular conduction delay (IVCD) with QRS ≥120 msec, left branch bundle block (LBBB), right branch bundle block (RBBB), Wolf-Parkinson- White syndrome (WPW), left anterior fascicular block (LAFB), left posterior fascicular block (LPFB), or other conduction abnormality that in the opinion of the investigator would preclude safe participation in this study.
* Females who are pregnant or lactating
* Known hypersensitivity to pegfilgrastim or filgrastim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed 2 cycles of treatment are considered having completed study.
Groups:
- 0.125 mg/m²/Day LY: 0.125 milligrams per meter square per day (mg/m²/day) LY2523355 (LY) was administered as an intravenous (IV) infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until progressive disease (PD), unacceptable toxicity or other withdrawal criterion is met.
- 0.25 mg/m²/Day LY: 0.25 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 0.5 mg/m²/Day LY: 0.5 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 1.0 mg/m²/Day LY: 1.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 2.0 mg/m²/Day LY: 2.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 4.0 mg/m²/Day LY: 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 5.0 mg/m²/Day LY: 5.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 6.0 mg/m²/Day LY: 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 4.0 mg/m²/Day LY + 6 mg PEG: 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles.
  6 milligrams (mg) pegfilgrastim (PEG) was administered subcutaneously (SC) on Day 4 of each 21-day cycle for at least 2 cycles and for any subsequent cycles of LY2523355 received.
  Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 6.0 mg/m²/Day LY + 6 mg PEG: 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles.
  6 mg pegfilgrastim was administered SC on Day 4 of each 21-day cycle for at least 2 cycles and for any subsequent cycles of LY2523355 received.
  Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 7.0 mg/m²/Day LY + 6 mg PEG: 7.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles.
  6 mg pegfilgrastim was administered SC on Day 4 of each 21-day cycle for at least 2 cycles and for any subsequent cycles of LY2523355 received.
  Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
Period: Overall Study
Arm/Group | 0.125 mg/m²/Day LY | 0.25 mg/m²/Day LY | 0.5 mg/m²/Day LY | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 4.0 mg/m²/Day LY + 6 mg PEG | 6.0 mg/m²/Day LY + 6 mg PEG | 7.0 mg/m²/Day LY + 6 mg PEG
Started | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3
Received at Least 1 Dose of Study Drug | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3
Completed | 0 | 0 | 1 | 1 | 1 | 9 | 4 | 2 | 2 | 11 | 1
Not Completed | 1 | 1 | 0 | 2 | 2 | 4 | 1 | 1 | 1 | 7 | 2
Not completed — Progressive Disease | 1 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 5 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.125 mg/m²/Day LY | 0.25 mg/m²/Day LY | 0.5 mg/m²/Day LY | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 4.0 mg/m²/Day LY + 6 mg PEG | 6.0 mg/m²/Day LY + 6 mg PEG | 7.0 mg/m²/Day LY + 6 mg PEG | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.01 (NA) — N of 1, no standard deviation | 71.20 (NA) — N of 1, no standard deviation | 52.37 (NA) — N of 1, no standard deviation | 60.78 (12.84) | 61.30 (13.91) | 59.79 (8.75) | 63.38 (12.50) | 67.26 (5.88) | 66.97 (17.19) | 56.82 (12.09) | 60.13 (0.49) | 60.27 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 3 | 3 | 9 | 3 | 1 | 3 | 12 | 2 | 37
  Male | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 2 | 0 | 6 | 1 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 9
  Caucasian | 0 | 0 | 1 | 3 | 2 | 10 | 5 | 3 | 2 | 10 | 2 | 38
  East Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hispanic | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 5
  Native American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3 | 54

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies
Description: Recommended Phase 2 dose was determined by the maximum tolerated dose (MTD). The MTD was defined as the dose that caused <1/3 of all participants treated with the study drug to experience a dose-limiting toxicity (DLT). A DLT was defined as an adverse event (AE) occurring during Cycle 1 that fulfilled 1 of the following criteria: Any Common Terminology Criteria for Adverse Events (CTCAE), version (v) 3.0 Grade ≥3 nonhematological toxicity possibly or likely related to the study drug (except for nausea/vomiting/diarrhea without maximal symptomatic/prophylactic treatment); any CTCAE v 3.0 Grade ≥3 thrombocytopenia with bleeding; any CTCAE v3.0 Grade 4 hematological toxicity of >5 days duration; any febrile neutropenia.
Time Frame: Baseline, daily up to 21 days in Cycle 1
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: mg/m²/day
Groups:
- LY2523355: 0.125 to 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle)
- LY2523355 + Pegfilgrastim: 4.0 to 7.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 with 6 mg pegfilgrastim administered SC on Day 4 of Cycle 1 (21-day Cycle).
Arm/Group | LY2523355 | LY2523355 + Pegfilgrastim
Number analyzed (Participants) | 30 | 24
mg/m²/day | 4.0 | 6.0

2. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Adverse events (AEs) were considered clinically significant effects. Data presented are the number of participants who experienced serious AEs (SAEs), other non-serious AEs and deaths during the study, including the 30-day follow-up. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion including 30-day follow-up up to 647 days,any AE reported
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 0.125 mg/m²/Day LY: 0.125 mg/m²/day LY2523355 (LY) was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles. Participants could continue on study drug until PD, unacceptable toxicity or other withdrawal criterion is met.
- 4.0 mg/m²/Day LY + 6 mg PEG: 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of each 21-day cycle for at least 2 cycles.
  6 mg pegfilgrastim (PEG) was administered subcutaneously (SC) on Day 4 of each 21-day cycle for at least 2 cycles and for any subsequent cycles of LY2523355 received.
  Participants could continue on study drug until PD unacceptable toxicity or other withdrawal criterion is met.
Arm/Group | 0.125 mg/m²/Day LY | 0.25 mg/m²/Day LY | 0.5 mg/m²/Day LY | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 4.0 mg/m²/Day LY + 6 mg PEG | 6.0 mg/m²/Day LY + 6 mg PEG | 7.0 mg/m²/Day LY + 6 mg PEG
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3
Participants
  SAEs | 0 | 0 | 0 | 1 | 0 | 5 | 3 | 3 | 0 | 11 | 3
  AEs | 1 | 1 | 0 | 2 | 3 | 13 | 5 | 3 | 3 | 18 | 3
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY2523355 Following A Single Dose
Description: Cmax following a single dose of LY2523355 at each dose level in the presence or absence of pegfilgrastim.
Time Frame: Cycle 1 Day 1(21-day cycle):End of infusion (EOI), Day 2: Predose, EOI, Day 3: Predose, EOI, between 1-2 hour EOI, Day 4: anytime, Day 8:anytime, Day 9: anytime, Day 10: anytime
Population: All enrolled participants who received 1 dose of LY2523355 on Day 1 of Cycle 1 with evaluable pharmacokinetic data to enable determination of the LY2523355 plasma Cmax on Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 1.0 mg/m²/Day LY: 1.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
- 2.0 mg/m²/Day LY: 2.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
- 4.0 mg/m²/Day LY: 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
- 5.0 mg/m²/Day LY: 5.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
- 6.0 mg/m²/Day LY: 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
- 7.0 mg/m²/Day LY: 7.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Day 1 of Cycle 1 (21-day cycle).
Arm/Group | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 7.0 mg/m²/Day LY
Number analyzed (Participants) | 3 | 3 | 16 | 5 | 21 | 3
nanograms/milliliter (ng/mL) | 32.6 (36) | 61.7 (10) | 120 (40) | 127 (28) | 168 (39) | 222 (33)

4. Secondary Outcome: Pharmacokinetics: Plasma Cmax of LY2523355 Following Multiple Doses
Description: Cmax following multiple doses of LY2523355 at each dose level in the presence or absence of pegfilgrastim.
Time Frame: Cycle 1, Day 3(21-day cycle): End of infusion
Population: All enrolled participants who received more than 1 dose of LY2523355 and had evaluable pharmacokinetic data to enable determination of the LY2523355 Cmax on Day 3 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 1.0 mg/m²/Day LY: 1.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle).
- 2.0 mg/m²/Day LY: 2.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle).
- 4.0 mg/m²/Day LY: 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle) or 4.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 with 6 mg pegfilgrastim administered SC on Day 4 of Cycle 1 (21-day cycle).
- 5.0 mg/m²/Day LY: 5.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle).
- 6.0 mg/m²/Day LY: 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 of Cycle 1 (21-day cycle) or 6.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 with 6 mg pegfilgrastim administered SC on Day 4 of Cycle 1 (21-day cycle).
- 7.0 mg/m²/Day LY: 7.0 mg/m²/day LY2523355 was administered as an IV infusion over 1 hour on Days 1, 2 and 3 with 6 mg pegfilgrastim administered SC on Day 4 of Cycle 1 (21-day cycle).
Arm/Group | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 7.0 mg/m²/Day LY
Number analyzed (Participants) | 3 | 3 | 16 | 5 | 20 | 3
ng/mL | 29.8 (32) | 73.6 (47) | 126 (49) | 129 (34) | 193 (37) | 231 (23)

5. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY2523355 Following A Single Dose
Description: AUC(0-∞) following a single dose of LY2523355 at each dose level in the presence or absence of pegfilgrastim.
Time Frame: Cycle 1,Day 1(21-day cycle): End of infusion (EOI), Day 2: Predose, EOI, Day 3: Predose, EOI, between 1-2 hour EOI, Day 4: anytime, Day 8:anytime, Day 9: anytime, Day 10: anytime
Population: All enrolled participants who received 1 dose of LY2523355 on Day 1 of Cycle 1 with evaluable pharmacokinetic data to enable calculation of the LY2523355 AUC(0-∞) on Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 7.0 mg/m²/Day LY
Number analyzed (Participants) | 3 | 3 | 16 | 5 | 21 | 3
nanograms*hour/milliliter (ng*h/mL) | 81.8 (33) | 159 (21) | 324 (41) | 379 (23) | 443 (40) | 642 (50)

6. Secondary Outcome: Pharmacokinetics: AUC(0-∞) of LY2523355 Following Multiple Doses
Description: AUC(0-∞) following multiple doses of LY2523355 at each dose level in the presence or absence of pegfilgrastim.
Time Frame: Cycle 1, Day 3(21-day cycle): End of infusion
Population: All enrolled participants who received more than 1 dose of LY2523355 and had evaluable pharmacokinetic data to enable calculation of the LY2523355 AUC(0-∞) on Day 3 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 7.0 mg/m²/Day LY
Number analyzed (Participants) | 3 | 3 | 16 | 5 | 20 | 3
ng*h/mL | 109 (19) | 220 (30) | 484 (46) | 593 (45) | 649 (52) | 1090 (54)

7. Secondary Outcome: Number of Participants With Tumor Response
Description: Data presented are the number of participants with a confirmed complete response (CR) or partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR is the disappearance of all target and non-target lesions. PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesions.
Time Frame: Baseline to measured disease progression or discontinuation up to 617 days
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.125 mg/m²/Day LY | 0.25 mg/m²/Day LY | 0.5 mg/m²/Day LY | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 4.0 mg/m²/Day LY + 6 mg PEG | 6.0 mg/m²/Day LY + 6 mg PEG | 7.0 mg/m²/Day LY + 6 mg PEG
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 13 | 5 | 3 | 3 | 18 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | 0.125 mg/m²/Day LY | 0.25 mg/m²/Day LY | 0.5 mg/m²/Day LY | 1.0 mg/m²/Day LY | 2.0 mg/m²/Day LY | 4.0 mg/m²/Day LY | 4.0 mg/m²/Day LY + 6 mg PEG | 5.0 mg/m²/Day LY | 6.0 mg/m²/Day LY | 6.0 mg/m²/Day LY + 6 mg PEG | 7.0 mg/m²/Day LY + 6 mg PEG
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 1/3 | 0/3 | 5/13 | 0/3 | 3/5 | 3/3 | 11/18 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 2/3 | 3/3 | 13/13 | 3/3 | 5/5 | 3/3 | 18/18 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.125 mg/m²/Day LY (N=1) | 0.25 mg/m²/Day LY (N=1) | 0.5 mg/m²/Day LY (N=1) | 1.0 mg/m²/Day LY (N=3) | 2.0 mg/m²/Day LY (N=3) | 4.0 mg/m²/Day LY (N=13) | 4.0 mg/m²/Day LY + 6 mg PEG (N=3) | 5.0 mg/m²/Day LY (N=5) | 6.0 mg/m²/Day LY (N=3) | 6.0 mg/m²/Day LY + 6 mg PEG (N=18) | 7.0 mg/m²/Day LY + 6 mg PEG (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.125 mg/m²/Day LY (N=1) | 0.25 mg/m²/Day LY (N=1) | 0.5 mg/m²/Day LY (N=1) | 1.0 mg/m²/Day LY (N=3) | 2.0 mg/m²/Day LY (N=3) | 4.0 mg/m²/Day LY (N=13) | 4.0 mg/m²/Day LY + 6 mg PEG (N=3) | 5.0 mg/m²/Day LY (N=5) | 6.0 mg/m²/Day LY (N=3) | 6.0 mg/m²/Day LY + 6 mg PEG (N=18) | 7.0 mg/m²/Day LY + 6 mg PEG (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 6 (7) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 1 (2) | 5 (8) | 0 (0) | 5 (7) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 4 (8) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 0 (0) | 3 (4) | 0 (0) | 7 (9) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 7 (12) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 7 (7) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (8) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Platelet count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 0 (0)
Skin chapped (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days